CLINICAL TRIAL: NCT01566773
Title: A Randomized, Double Blind (Test Products and Placebo), Chronic Dosing (14 Days), Four Period, Eight Treatment, Placebo-Controlled, Incomplete Block, Cross Over, Multi Center Study to Assess Efficacy and Safety of Six Doses of PT001 in Patients With Moderate to Severe COPD, Compared With Spiriva® Handihaler® (Tiotropium Bromide, Open Label) as An Active Control
Brief Title: PT001 MDI Versus Spiriva® in Patients With Moderate to Severe COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT001003
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- PT001 MDI (Dose 1) (Experimental)
  Interventions: Drug: PT001 MDI
- PT001 MDI (Dose 2) (Experimental)
  Interventions: Drug: PT001 MDI
- PT001 MDI (Dose 3) (Experimental)
  Interventions: Drug: PT001 MDI
- PT001 MDI (Dose 4) (Experimental)
  Interventions: Drug: PT001 MDI
- PT001 MDI (Dose 5) (Experimental)
  Interventions: Drug: PT001 MDI
- PT001 MDI (Dose 6) (Experimental)
  Interventions: Drug: PT001 MDI
- PT001 Placebo MDI (Placebo Comparator)
  Interventions: Drug: PT001 Placebo MDI
- Spiriva® Handihaler® (Tiotropium Bromide) (Active Comparator)
  Interventions: Drug: Tiotropium Bromide

INTERVENTIONS:
Drug: PT001 MDI — Administered as two puffs BID for 14 days
  Arms: PT001 MDI (Dose 1); PT001 MDI (Dose 2); PT001 MDI (Dose 3); PT001 MDI (Dose 4); PT001 MDI (Dose 5); PT001 MDI (Dose 6)
Drug: Tiotropium Bromide — Taken as 1 capsule containing 18 µg of tiotropium via the Handihaler DPI
  Other Names: Spiriva® Handihaler®
  Arms: Spiriva® Handihaler® (Tiotropium Bromide)
Drug: PT001 Placebo MDI
  Arms: PT001 Placebo MDI

SUMMARY:
The overall objective of this study is to determine an optimal dose and dosing regimen of PT001 MDI for further evaluation in later stage studies.

DETAILED DESCRIPTION:
The primary objective of this study is to assess efficacy relative to placebo of GP MDI in subjects with moderate to severe chronic obstructive pulmonary disease (COPD) within the range of doses evaluated in this protocol. To this end, each dose of GP MDI will be compared to placebo with respect to the primary efficacy endpoint, FEV1 AUC0-12 relative to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* 40 - 80 years of age
* Clinical history of COPD with airflow limitation that is not fully reversible
* Females of non-child bearing potential or females of child bearing potential with negative pregnancy test; and acceptable contraceptive methods
* Current/former smokers with at least a 10 pack-year history of cigarette smoking
* A measured post- bronchodilator FEV1/FVC ratio of < or = 0.70
* A measured post- bronchodilator FEV1 > or = 750ml or 30% predicted and < or = 80% of predicted normal values
* Able to change COPD treatment as required by protocol

Exclusion Criteria:

* Women who are pregnant or lactating
* Primary diagnosis of asthma
* Alpha-1 antitrypsin deficiency as the cause of COPD
* Active pulmonary diseases
* Prior lung volume reduction surgery
* Abnormal chest X-ray (or CT scan) not due to the presence of COPD
* Hospitalized due to poorly controlled COPD within 3 months of Screening
* Clinically significant medical conditions that preclude participation in the study (e.g. clinically significant abnormal ECG, uncontrolled hypertension, glaucoma, symptomatic prostatic hypertrophy)
* Cancer that has not been in complete remission for at least 5 years
* Treatment with investigational study drug or participation in another clinical trial or study within the last 30 days or 5 half lives

Other inclusion/exclusion criteria as defined in the protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, MD, Study Director — Pearl Therapeutics, Inc.
Locations (10):
- United States (10):
  - Pearl Investigative Site, Fullerton, California
  - Pearl Investigative Site, Clearwater, Florida
  - Pearl Investigative Site, Panama City, Florida
  - Pearl Investigative Site, Tampa, Florida
  - Pearl Investigative Site, Winter Park, Florida
  - Pearl Investigative Site, Charlotte, North Carolina
  - Pearl Investigative Site, Medford, Oregon
  - Pearl Investigative Site, Spartanburg, South Carolina
  - Pearl Investigative Site, Longview, Texas
  - Pearl Investigative Site, Richmond, Virginia

REFERENCES:
- [Derived] Fabbri LM, Kerwin EM, Spangenthal S, Ferguson GT, Rodriguez-Roisin R, Pearle J, Sethi S, Orevillo C, Darken P, St Rose E, Fischer T, Golden M, Dwivedi S, Reisner C. Dose-response to inhaled glycopyrrolate delivered with a novel Co-Suspension Delivery Technology metered dose inhaler (MDI) in patients with moderate-to-severe COPD. Respir Res. 2016 Sep 2;17(1):109. doi: 10.1186/s12931-016-0426-4. PMID 27586537
- See also: protocol-pt001003_FINAL_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4161&filename=protocol-pt001003_FINAL_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 sites in the US from April 2012 to August 2012. Study participation maximum of 26 weeks.
Pre-assignment Details: A randomized, double-blind,chronic dosing, four-period, eight-treatment, placebo-controlled, incomplete block, crossover, multicenter study.
Period: Overall Study
Arm/Group | All Subjects
Started | 140
GP MDI 18 µg BID | 64
GP MDI 9 µg BID | 64
GP MDI 4.6 µg BID | 62
GP MDI 2.4 µg BID | 64
GP MDI 1.2 µg BID | 57
GP MDI 0.6 µg BID | 59
Placebo MDI | 62
Spiriva® Handihaler® | 62
Completed | 110
Not Completed | 30
Not completed — Protocol specified criteria | 4
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 9
Not completed — Administrative reason | 1
Not completed — Adverse Event | 10
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population: Subjects who randomized and received at least 1 dose of study drug, and had both baseline and post-baseline efficacy data for that treatment.
Groups:
- All Subjects: All Subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 75

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC0-12
Description: Forced expiratory volume in 1 second (FEV1) normalized area under the curve 0-12 hours (AUC0-12) following chronic dosing for 14 days.
Time Frame: Day 14 (-1 hr, -30 min, 15 min, 30 min, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 10 hr, 11.5 hr, 12 hr)
Population: MITT (Modified Intent to Treat) Population: Subjects who completed at least 2 treatment periods with minimally 2 hours post-dosing on Day 14 for each of the treatment periods.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Groups:
- GP MDI 18 µg BID: GP MDI 18 µg BID.
- GP MDI 9 µg BID: GP MDI 9 µg BID.
- GP MDI 4.6 µg BID: GP MDI 4.6 µg BID.
- GP MDI 2.4 µg BID: GP MDI 2.4 µg BID.
- GP MDI 1.2 µg BID: GP MDI 1.2 µg BID.
- GP MDI 0.6 µg BID: GP MDI 0.6 µg BID.
- Placebo MDI: Placebo MDI.
- Spiriva® Handihaler®: Spiriva® Handihaler® (Tiotropium Bromide).
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 58 | 59 | 60 | 53 | 54 | 52 | 55
Liter | 1.448 [1.405 to 1.491] | 1.416 [1.374 to 1.459] | 1.432 [1.389 to 1.474] | 1.416 [1.374 to 1.458] | 1.386 [1.342 to 1.430] | 1.353 [1.309 to 1.397] | 1.290 [1.246 to 1.335] | 1.514 [1.471 to 1.558]

2. Secondary Outcome: Peak Change From Baseline in FEV1
Description: Highest value of FEV1 post dose on day 1
Time Frame: Day 1
Population: MITT Population: Subjects who completed at least 2 treatment periods with minimally 2 hours post-dosing on Day 14 for each of the treatment periods.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 59 | 59 | 60 | 59 | 55 | 55 | 60 | 57
mL | 231 [191 to 272] | 226 [186 to 267] | 165 [125 to 205] | 170 [130 to 211] | 136 [95 to 177] | 107 [65 to 149] | 57 [17 to 97] | 270 [229 to 311]

3. Secondary Outcome: Time to Onset of Action (>10% Improvement in FEV1) on Day 1
Description: Time to Onset of Action (>10% Improvement in FEV1) on Day 1.
Time Frame: Day 1 (15 min, 30 min, 1 hr, 2 hrs, no onset within 2 hrs)
Population: as for outcome 2
Measure: Number; unit: % of participants
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 55 | 56 | 57 | 58 | 50 | 54 | 55 | 54
% of participants
  15 minutes | 29 | 30 | 14 | 21 | 18 | 7 | 4 | 39
  30 minutes | 22 | 11 | 9 | 16 | 12 | 9 | 7 | 15
  1 hour | 26 | 11 | 11 | 10 | 10 | 17 | 9 | 15
  2 hours | 0 | 16 | 11 | 7 | 10 | 7 | 2 | 11
  No onset within 2 hours | 24 | 32 | 56 | 47 | 50 | 59 | 78 | 20

4. Secondary Outcome: Percentage of Subjects Achieving at Least 12% Improvement in FEV1
Description: Percentage of subjects achieving at least 12% improvement in FEV1.
Time Frame: Day 1
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 56 | 58 | 60 | 52 | 56 | 56
Percentage of participants | 70 | 59 | 40 | 47 | 40 | 31 | 71

5. Secondary Outcome: Peak Change From Baseline in Inspiratory Capacity (IC)
Description: Peak change in Inspiratory Capacity (IC) mean of 1 and 2 hour post-dose assessments minus the baseline
Time Frame: Day 1 (1 hr and 2 hr post-dose )
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 59 | 59 | 61 | 60 | 55 | 54 | 60 | 56
mL | 234 [163 to 304] | 263 [193 to 333] | 151 [82 to 219] | 183 [113 to 252] | 126 [54 to 198] | 82 [9 to 155] | 80 [10 to 150] | 343 [271 to 414]

6. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1
Description: Change from baseline in morning pre-dose trough FEV1 (average of the 60 and 30-minute pre-dose values on Treatment Day 7 minus the baseline)
Time Frame: Day 7 (average of the 60 and 30-minute pre-dose values on Treatment Day 7 minus the baseline)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 59 | 60 | 60 | 55 | 55 | 58 | 57
mL | 88 [48 to 128] | 90 [50 to 129] | 109 [70 to 149] | 96 [57 to 135] | 43 [2 to 84] | 23 [-18 to 64] | 10 [-29 to 50] | 156 [116 to 196]

7. Secondary Outcome: Peak Change From Baseline in FEV1
Description: Peak change from baseline in FEV1 (defined as the change at the highest value of FEV1 post-dose minus the baseline)
Time Frame: Day 7
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 59 | 59 | 59 | 55 | 54 | 58 | 57
mL | 286 [239 to 333] | 269 [223 to 316] | 266 [220 to 313] | 235 [189 to 282] | 225 [178 to 273] | 166 [118 to 214] | 114 [67 to 161] | 366 [318 to 413]

8. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough Inspiratory Capacity (IC)
Description: Change from baseline in morning pre-dose trough IC (average of the 60 and 30-minute pre-dose assessments minus the baseline)
Time Frame: Day 7
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 59 | 60 | 60 | 55 | 54 | 58 | 56
mL | 137 [75 to 198] | 57 [-4 to 118] | 101 [40 to 162] | 142 [81 to 203] | 73 [10 to 137] | 54 [-10 to 118] | 62 [1 to 124] | 184 [121 to 247]

9. Secondary Outcome: Peak Change From Baseline in IC
Description: Peak change from baseline in IC (mean of 1 hr and 2 hr post-dose assessments)
Time Frame: Day 7 (mean of 1 hr and 2 hr post-dose assessments)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 59 | 60 | 60 | 55 | 54 | 58 | 56
mL | 302 [227 to 377] | 234 [160 to 309] | 254 [180 to 328] | 312 [238 to 386] | 195 [118 to 272] | 159 [82 to 236] | 99 [24 to 174] | 390 [314 to 466]

10. Secondary Outcome: Change From Baseline in Mean Morning Pre-dose Daily PEFR
Description: Change from baseline in mean morning pre-dose daily PEFR (peak expiratory flow rate) taken by subjects and recorded in subject diaries, up through Diary Day 7 of each treatment period (excluding reading taken pre-dose on Visit 2 [Treatment Day 1])
Time Frame: Day 7 (60 minutes pre-dose, 30 minutes pre-dose)
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 58 | 59 | 59 | 55 | 55 | 59 | 56
L/min | 8.0 [1.1 to 15.0] | 3.2 [-3.7 to 10.2] | 0.2 [-6.7 to 7.1] | 2.4 [-4.5 to 9.3] | -2.4 [-9.5 to 4.6] | -2.5 [-9.5 to 4.6] | -7.2 [-14.1 to -0.3] | 12.7 [5.6 to 19.7]

11. Secondary Outcome: Change From Baseline in Morning Post-dose Daily PEFR
Description: Change from baseline in morning post-dose daily PEFR (peak expiratory flow rate) taken by subjects and recorded in subject diaries, up through Diary Day 7 of each treatment period (excluding reading taken pre-dose on Visit 2 [Treatment Day 1])
Time Frame: Day 7 (30 minutes post-dose)
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 58 | 59 | 59 | 55 | 55 | 59 | 56
L/min | 32.3 [24.8 to 39.8] | 23.9 [16.5 to 31.4] | 17.2 [9.8 to 24.6] | 18.3 [10.8 to 25.7] | 14.3 [6.6 to 21.9] | 13.7 [6.0 to 21.3] | 4.5 [-2.9 to 12.0] | 38.0 [30.4 to 45.6]

12. Secondary Outcome: Change From Baseline in Mean Evening Pre-dose PEFR
Description: Change from baseline in mean evening pre-dose daily peak flow readings taken by subjects and recorded in subject diaries, up through Diary Day 7 of each treatment period (subjects taking Spiriva performed a single evening assessment)
Time Frame: Day 7
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI
Number analyzed (Participants) | 58 | 58 | 59 | 59 | 55 | 55 | 59
L/min | 15.8 [8.6 to 22.9] | 12.6 [5.6 to 19.6] | 4.7 [-2.3 to 11.7] | 11.2 [4.2 to 18.3] | 7.5 [0.2 to 14.7] | 5.9 [-1.3 to 13.1] | 3.3 [-3.8 to 10.4]

13. Secondary Outcome: Change From Baseline in Mean Evening Post-dose PEFR
Description: Change from baseline in mean evening post-dose daily peak flow readings taken by subjects and recorded in subject diaries, up through Diary Day 7 of each treatment period (subjects taking Spiriva performed a single evening assessment)
Time Frame: Day 7
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Groups:
- Spiriva Respimat: Spiriva Respimat 18 µg
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva Respimat
Number analyzed (Participants) | 58 | 58 | 59 | 59 | 55 | 55 | 59 | 55
L/min | 42.2 [34.2 to 50.2] | 30.3 [22.4 to 38.3] | 21.6 [13.7 to 29.5] | 24.3 [16.3 to 32.3] | 20.2 [12.1 to 28.3] | 22.1 [14.0 to 30.2] | 11.0 [3.1 to 19.0] | 35.6 [27.4 to 43.7]

14. Secondary Outcome: Mean Number of Puffs of Rescue Medication
Description: Mean number of puffs of rescue medication recorded in subject diaries during each treatment period and by treatment and numbers of days treated
Time Frame: Day 7
Population: MITT Population
Measure: Mean (95% Confidence Interval); unit: Puffs
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 59 | 59 | 61 | 60 | 55 | 55 | 60 | 58
Puffs | 0.9 [0.60 to 1.37] | 1.3 [0.88 to 1.89] | 1.2 [0.85 to 1.71] | 1.2 [0.82 to 1.58] | 1.5 [1.03 to 1.99] | 1.6 [1.12 to 2.19] | 2.0 [1.46 to 2.66] | 0.9 [0.63 to 1.28]

15. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1
Description: Change from baseline in morning pre-dose trough FEV1 (average of the 60 and 30-minute pre-dose values on Treatment Day 14 minus the baseline)
Time Frame: Day 14 (average of the 60 and 30-minute pre-dose values on Treatment Day 14 minus the baseline)
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 59 | 60 | 59 | 55 | 55 | 56 | 57
mL | 89 [47 to 132] | 80 [38 to 122] | 67 [26 to 109] | 77 [35 to 118] | 68 [25 to 111] | 29 [-14 to 72] | -8 [-50 to 35] | 126 [84 to 168]

16. Secondary Outcome: Peak Change From Baseline in FEV1
Description: Peak change from baseline in FEV1 (defined as the change at the highest value of FEV1 post-dose minus the baseline)
Time Frame: Day 14
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 59 | 60 | 60 | 54 | 54 | 54 | 57
mL | 288 [236 to 339] | 288 [237 to 340] | 287 [236 to 338] | 261 [210 to 312] | 246 [193 to 299] | 188 [135 to 241] | 130 [77 to 183] | 361 [309 to 413]

17. Secondary Outcome: Change From Baseline for Mean Morning Pre-dose Trough IC
Description: Change from baseline for mean morning pre-dose trough IC (average of the 60 and 30-minute pre-dose assessments minus the baseline)
Time Frame: Day 14 (average of the 60 and 30-minute pre-dose assessments minus the baseline)
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 59 | 60 | 60 | 55 | 54 | 56 | 56
mL | 94 [32 to 156] | 45 [-16 to 106] | 64 [3 to 124] | 104 [43 to 165] | 69 [6 to 132] | 34 [-30 to 97] | 9 [-54 to 71] | 138 [76 to 201]

18. Secondary Outcome: Peak Change From Baseline in IC
Description: Peak change from baseline in IC (mean of 1 and 2 hour post-dose assessments minus the baseline)
Time Frame: Day 14 (mean of 1 and 2 hour post-dose assessments minus the baseline)
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 59 | 60 | 60 | 54 | 54 | 56 | 56
mL | 280 [197 to 363] | 259 [177 to 341] | 288 [206 to 370] | 226 [145 to 308] | 261 [176 to 346] | 172 [87 to 256] | 77 [-6 to 161] | 284 [200 to 368]

19. Secondary Outcome: Change From Baseline in 12-hour Post-dose Trough FEV1
Description: 12-hour post-dose trough FEV1 was defined as the mean of the FEV1 assessments taken at 11.5 and 12 hours post-dose minus the baseline
Time Frame: Day 14 (Baseline, 11.5 and 12 hours post dose)
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 58 | 59 | 60 | 53 | 55 | 54 | 56
mL | 116 [69 to 163] | 69 [22 to 117] | 99 [52 to 145] | 112 [65 to 158] | 66 [17 to 115] | 55 [7 to 104] | 1 [-48 to 49] | 164 [116 to 211]

20. Secondary Outcome: Change From Baseline in Mean Morning Pre-dose Daily PEFR
Description: Change from baseline in mean morning pre-dose daily peak flow readings taken by subjects and recorded in subject diaries during each treatment period for subjects with more than 7 days of diary data (mean reading excluded reading taken pre-dose on Visit 2 [Treatment 1 Day 1]
Time Frame: Baseline, Treatment Day 1 and every day, to the end of the 14-Day Treatment period before dosing, values were averaged for the end of treatment value (all subjects with diary data after Diary day 7)
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 57 | 58 | 59 | 59 | 55 | 55 | 58 | 56
L/min | 8.6 [2.1 to 15.1] | 6.2 [-0.3 to 12.8] | 2.0 [-4.5 to 8.5] | 4.4 [-2.1 to 10.9] | 0.3 [-6.4 to 6.9] | -0.5 [-7.1 to 6.2] | -6.3 [-12.7 to 0.2] | 14.8 [8.2 to 21.4]

21. Secondary Outcome: Change From Baseline in Mean Morning Post-dose Daily PEFR
Description: Change from baseline in mean morning post-dose daily peak flow readings taken by subjects and recorded in subject diaries during each treatment period for subjects with more than 7 days of diary data (mean reading excluded reading taken pre-dose on Visit 2 [Treatment 1 Day 1]
Time Frame: Baseline, Treatment Day 1 and every day, to the end of the 14-Day Treatment period 30 minutes post dosing, values were averaged for the end of treatment value (all subjects with diary data after Diary day 7)
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 57 | 58 | 59 | 59 | 55 | 55 | 58 | 56
L/min | 33.5 [25.8 to 40.4] | 26.7 [19.4 to 33.9] | 20.2 [13.0 to 27.4] | 20.3 [13.1 to 27.5] | 14.8 [7.5 to 22.2] | 14.3 [6.9 to 21.7] | 5.3 [-1.9 to 12.5] | 39.8 [32.5 to 47.1]

22. Secondary Outcome: Change From Baseline in Mean Evening Pre-dose Daily PEFR
Description: Change from baseline in mean evening pre-dose daily peak flow readings taken by subjects and recorded in subject diaries during each treatment period for subjects with more than 7 days of diary data (subjects taking Spiriva performed a single evening assessment)
Time Frame: Treatment Day 1 to the end of the 14-Day Treatment, values were averaged for the end of treatment value (all subjects with diary data after Diary day 7)
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI
Number analyzed (Participants) | 57 | 58 | 59 | 59 | 55 | 55 | 58
L/min | 15.7 [8.8 to 22.5] | 14.9 [8.1 to 21.7] | 7.2 [0.5 to 13.9] | 11.7 [4.9 to 18.5] | 5.0 [-1.9 to 12.0] | 6.9 [-0.0 to 13.8] | 5.7 [-1.1 to 12.6]

23. Secondary Outcome: Change From Baseline in Mean Evening Post-dose Daily PEFR
Description: Change from baseline in mean evening post-dose daily peak flow readings taken by subjects and recorded in subject diaries during each treatment period for subjects with more than 7 days of diary data (subjects taking Spiriva performed a single evening assessment)
Time Frame: Through the end of the 14-Day Treatment
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 57 | 58 | 59 | 59 | 55 | 55 | 58 | 56
L/min | 41.4 [33.6 to 49.2] | 32.7 [24.9 to 40.5] | 24.7 [16.9 to 32.4] | 27.0 [19.3 to 34.8] | 19.4 [11.5 to 27.3] | 22.7 [14.8 to 30.6] | 13.5 [5.8 to 21.3] | 35.9 [28.1 to 43.8]

24. Secondary Outcome: Mean Number of Puffs of Rescue Medication (End of Treatment)
Description: as for outcome 14
Time Frame: Day 14 (End of treatment)
Population: MITT Population
Measure: Mean (95% Confidence Interval); unit: Puffs
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 59 | 59 | 61 | 60 | 55 | 55 | 68 | 58
Puffs | 0.85 [0.56 to 1.28] | 1.25 [0.83 to 1.81] | 1.19 [0.83 to 1.66] | 1.11 [0.79 to 1.51] | 1.43 [1.02 to 1.95] | 1.57 [1.12 to 2.15] | 1.92 [1.39 to 2.56] | 0.87 [0.60 to 1.29]

25. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 (mL) Averaging Treatment Day 7 and Day 14
Description: Change from Baseline in Morning Pre-dose Trough FEV1 (mL) Averaging Treatment Day 7 and Day 14
Time Frame: Day 1 through Day 14
Population: MITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva® Handihaler®
Number analyzed (Participants) | 58 | 59 | 60 | 59 | 55 | 55 | 56 | 57
Liter | 0.088 [0.053 to 0.123] | 0.087 [0.052 to 0.121] | 0.090 [0.056 to 0.124] | 0.086 [0.052 to 0.120] | 0.056 [0.021 to 0.091] | 0.023 [-0.013 to 0.058] | 0.001 [-0.034 to 0.036] | 0.141 [0.107 to 0.176]

ADVERSE EVENTS:
Time Frame: All of the adverse events (AEs) reported during the study were captured after signing informed consent through the 7-14 day follow up period.
Groups:
- Spiriva 18 µg: Spiriva 18 µg
Arm/Group | GP MDI 18 µg BID | GP MDI 9 µg BID | GP MDI 4.6 µg BID | GP MDI 2.4 µg BID | GP MDI 1.2 µg BID | GP MDI 0.6 µg BID | Placebo MDI | Spiriva 18 µg
Serious Adverse Events (participants affected / at risk) | 0/64 | 1/64 | 0/62 | 1/64 | 0/57 | 1/59 | 1/62 | 1/62
Other Adverse Events (participants affected / at risk) | 2/64 | 3/64 | 3/62 | 6/64 | 3/57 | 4/59 | 3/62 | 6/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP MDI 18 µg BID (N=64) | GP MDI 9 µg BID (N=64) | GP MDI 4.6 µg BID (N=62) | GP MDI 2.4 µg BID (N=64) | GP MDI 1.2 µg BID (N=57) | GP MDI 0.6 µg BID (N=59) | Placebo MDI (N=62) | Spiriva 18 µg (N=62)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP MDI 18 µg BID (N=64) | GP MDI 9 µg BID (N=64) | GP MDI 4.6 µg BID (N=62) | GP MDI 2.4 µg BID (N=64) | GP MDI 1.2 µg BID (N=57) | GP MDI 0.6 µg BID (N=59) | Placebo MDI (N=62) | Spiriva 18 µg (N=62)
Dry mouth (Gastrointestinal disorders) | 2 (4) | 3 (3) | 3 (3) | 6 (7) | 3 (3) | 4 (5) | 3 (3) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.